CLINICAL TRIAL: NCT03045341
Title: Behavioral and Pharmacologic Treatment of Binge Eating and Obesity
Brief Title: Behavioral and Pharmacologic Treatment of Binge Eating and Obesity: Acute Treatment
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1506016065-A; R01DK049587 (NIH)
Record Dates: First submitted 2017-02-03; First posted 2017-02-07 (Estimated); Results first posted 2022-12-20 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Binge-eating Disorder; Obesity
MeSH Terms: conditions — Binge-Eating Disorder; Obesity | interventions — Naltrexone-Bupropion combination; bupropion hydrochloride, naltrexone hydrochoride drug combination; Counseling

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BWL + NB medication (Experimental): Participants randomly assigned to this arm will receive 16 weeks of Behavioral Weight Loss (BWL) counseling and NB medication. NB medication will combine naltrexone sustained-release (SR, 32 mg/day) combined with bupropion SR (360 mg/day) taken daily in pill form.
  Interventions: Drug: NB medication (Naltrexone Bupropion combination); Behavioral: Behavioral Weight Loss (BWL) counseling
- BWL + Placebo (Experimental): Participants randomly assigned to this arm will receive 16 weeks of Behavioral Weight Loss (BWL) counseling and placebo. Placebo will be inactive and taken daily in pill form.
  Interventions: Behavioral: Behavioral Weight Loss (BWL) counseling; Other: Placebo
- NB medication (Experimental): Participants randomly assigned to this arm will receive 16 weeks of NB medication. NB medication will combine naltrexone sustained-release (SR, 32 mg/day) combined with bupropion SR (360 mg/day) taken daily in pill form.
  Interventions: Drug: NB medication (Naltrexone Bupropion combination)
- Placebo (Placebo Comparator): Participants randomly assigned to this arm will receive 16 weeks of placebo. Placebo will be inactive and taken daily in pill form.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: NB medication (Naltrexone Bupropion combination) — NB medication
  Other Names: Contrave
  Arms: BWL + NB medication; NB medication
Behavioral: Behavioral Weight Loss (BWL) counseling — BWL counseling
  Arms: BWL + NB medication; BWL + Placebo
Other: Placebo — Placebo
  Arms: BWL + Placebo; Placebo

SUMMARY:
This study will test the effectiveness and relative efficacy of behavioral and pharmacologic treatments, alone and in combination, for the treatment of binge eating disorder (BED) in patients with obesity. This is an acute treatment comparing behavioral weight loss alone or in combination with naltrexone/bupropion medication.

DETAILED DESCRIPTION:
Binge eating disorder (BED), the most prevalent formal eating disorder, is associated strongly with obesity and bio-psychosocial impairment. Improved treatments for obese patients with BED are needed that can produce sustained clinical outcomes and promote weight loss. This study (acute treatment stage) aims to test the effectiveness of behavioral weight loss (BWL) and pharmacological treatment with Naltrexone/Bupropion (NB; a recently FDA-approved anti-obesity combination medication), alone and in combination, for the treatment of BED in patients with obesity. The acute treatment stage stage RCT will provide new findings regarding the effectiveness of NB medication and whether this specific combination of BWL and NB medication is effective for patients with obesity and BED. N=160 patients with BED and obesity will be randomly assigned (double-blind) in a balanced factorial (2 X 2) design trial, to one of four 16-week interventions: BWL+NB, BWL+Placebo, NB, or Placebo. This study will produce important new information about the relative efficacy of BWL and this recently FDA-approved anti-obesity (NB medicine), alone and in combination, for BED in patients with obesity.

ELIGIBILITY:
Inclusion Criteria:

* Binge eating disorder (full criteria as described in the American Psychiatric Association Diagnostic and Statistical Manual of Mental Disorders, 5th edition)
* BMI 27-30 with a controlled obesity-related co-morbidity; or BMI ≥ 30 and <50;
* Available for the duration of the treatment and follow-up (20 months);
* Read, comprehend, and write English at a sufficient level to complete study-related materials;
* Able to travel to study location (New Haven, CT) for weekly visits.

Exclusion Criteria:

* Currently taking anti-depressant medications;
* Currently taking opioid pain medications or drugs;
* Currently taking medications that influence eating/weight;
* History of seizures;
* Current substance use disorder or other severe psychiatric disturbance (e.g., suicidality);
* Past or current anorexia nervosa, bulimia nervosa;
* Pregnant or breastfeeding;
* Medical status judged by study physician as contraindication.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2021-07-23 (Actual); Study Completion 2022-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Grilo, PhD, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Grilo CM, Lydecker JA, Fineberg SK, Moreno JO, Ivezaj V, Gueorguieva R. Naltrexone-Bupropion and Behavior Therapy, Alone and Combined, for Binge-Eating Disorder: Randomized Double-Blind Placebo-Controlled Trial. Am J Psychiatry. 2022 Dec 1;179(12):927-937. doi: 10.1176/appi.ajp.20220267. Epub 2022 Oct 26. PMID 36285406

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | NB Medication | BWL + Placebo | BWL + NB Medication
Started | 34 | 32 | 35 | 35
Completed | 29 | 27 | 27 | 29
Not Completed | 5 | 5 | 8 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | NB Medication | BWL + Placebo | BWL + NB Medication | Total
Number analyzed (Participants) | 34 | 32 | 35 | 35 | 136
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.94 (12.57) | 46.03 (11.95) | 46.00 (11.87) | 46.99 (12.98) | 46.50 (12.23)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 6 | 5 | 5 | 6 | 22
  Female | 28 | 26 | 28 | 29 | 111
  Other | 0 | 1 | 2 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 7 | 5 | 4 | 20
  Not Hispanic or Latino | 30 | 25 | 30 | 31 | 116
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 1 | 0 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 3 | 8 | 4 | 18
  White | 26 | 25 | 26 | 29 | 106
  More than one race | 2 | 3 | 1 | 1 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Sexual Orientation [Count of Participants; unit: Participants]
  Heterosexual | 30 | 29 | 33 | 33 | 125
  Gay or Lesbian | 2 | 0 | 1 | 1 | 4
  Bisexual | 1 | 2 | 0 | 1 | 4
  Other | 1 | 1 | 1 | 0 | 3
Education [Count of Participants; unit: Participants]
  High School | 7 | 5 | 4 | 5 | 21
  Some College | 9 | 6 | 14 | 11 | 40
  College | 10 | 7 | 5 | 10 | 32
  More than College | 8 | 14 | 12 | 9 | 43

OUTCOME MEASURES:

1. Primary Outcome: Binge Eating Frequency (Continuous)
Description: Binge eating will be assessed by interview and self-report and the primary outcome is frequency. Frequency will be defined continuously (analyzed dimensionally).
Time Frame: Post-treatment (4 months)
Measure: Mean (Standard Deviation); unit: binge-eating episodes per month
Arm/Group | Placebo | NB Medication | BWL + Placebo | BWL + NB Medication
Number analyzed (Participants) | 29 | 27 | 27 | 29
binge-eating episodes per month | 9.90 (20.31) | 7.63 (9.77) | 3.30 (5.28) | 1.97 (4.87)
Statistical Analysis 1: Comparison: Placebo vs NB Medication vs BWL + Placebo vs BWL + NB Medication; BWL versus no BWL; Test type: Superiority — Analyses used all available data; p = 0.0001, Mixed Models Analysis; Analyses to compare treatments were all intent-to-treat. Analyses were performed for all randomized patients who attended the first treatment session
Statistical Analysis 2: Comparison: Placebo vs NB Medication vs BWL + Placebo vs BWL + NB Medication; NB versus placebo; Test type: Superiority — Analyses used all available data; p = 0.58, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]

2. Primary Outcome: Body Mass Index (Percent Weight Loss)
Description: BMI is calculated using measured height and weight. Percent weight loss, where negative values represent proportional weight loss, is calculated as the difference between weight at post-treatment and baseline weight, divided by baseline weight. By definition, all participants have 0% weight loss at baseline.
Time Frame: Post-treatment (4 months)
Population: Analyses used all available data.
Measure: Mean (Standard Deviation); unit: percentage of baseline weight
Arm/Group | Placebo | NB Medication | BWL + Placebo | BWL + NB Medication
Number analyzed (Participants) | 29 | 26 | 26 | 29
percentage of baseline weight | 1.05 (4.26) | -2.11 (5.41) | -4.42 (5.70) | -5.71 (5.85)
Statistical Analysis 1: Comparison: Placebo vs NB Medication vs BWL + Placebo vs BWL + NB Medication; BWL versus no BWL; Test type: Superiority — Analyses used all available data; p = 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs NB Medication vs BWL + Placebo vs BWL + NB Medication; NB versus placebo; Test type: Superiority — Analyses used all available data; p = 0.63, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Number of Participants Meeting Response Criteria
Description: Binge eating frequency will be assessed by interview and self-report. Frequency is defined categorically (response to treatment or non-response to treatment). Response to treatment is defined as a 65% reduction in binge eating frequency in past month, compared to baseline.
Time Frame: Post-treatment (4 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | NB Medication | BWL + Placebo | BWL + NB Medication
Number analyzed (Participants) | 29 | 27 | 26 | 29
Participants | 14 | 14 | 20 | 25
Statistical Analysis 1: Comparison: Placebo vs NB Medication vs BWL + Placebo vs BWL + NB Medication; Analyses used all available data; Test type: Superiority; p = .004, Chi-squared

ADVERSE EVENTS:
Time Frame: Month 1
Description: Participants were interviewed by research clinicians. For non-serious adverse events that were listed as >5% on the package insert for "Contrave" (naltrexone HCl/ bupropion HCl), we provide the total participants [all available data] who reported the adverse event at month 1.
Arm/Group | Placebo | NB Medication | BWL + Placebo | BWL + NB Medication
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/27 | 0/29 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/27 | 1/29 | 0/31
Other Adverse Events (participants affected / at risk) | 18/31 | 24/27 | 20/29 | 24/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=31) | NB Medication (N=27) | BWL + Placebo (N=29) | BWL + NB Medication (N=31)
Hypertensive Crisis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=31) | NB Medication (N=27) | BWL + Placebo (N=29) | BWL + NB Medication (N=31)
Anxiety (Psychiatric disorders) | 4 | 3 | 2 | 3
Constipation (Gastrointestinal disorders) | 6 | 11 | 7 | 8
Diarrhea (Gastrointestinal disorders) | 9 | 3 | 3 | 4
Dizziness (General disorders) | 1 | 12 | 3 | 5
Dry Mouth (General disorders) | 4 | 16 | 4 | 11
Headache (General disorders) | 7 | 13 | 9 | 11
Insomnia (General disorders) | 7 | 11 | 3 | 6
Nausea (Gastrointestinal disorders) | 5 | 13 | 3 | 8
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-28): https://cdn.clinicaltrials.gov/large-docs/41/NCT03045341/Prot_SAP_000.pdf